CLINICAL TRIAL: NCT04882397
Title: Immidate Effect of Instrument Assited Soft Tissue Mobilization Technique on Pain and Joint Position Sense in Individuals With Chronic Neck Pain
Brief Title: Immidate Effect of Instrument Assited Soft Tissue Mobilization Technique on Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KaratayUH3
Record Dates: First submitted 2021-05-08; First posted 2021-05-12 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2021-05

CONDITIONS: Neck Pain
Keywords: Joint Position Sense; Soft Tissue; Mobilization; Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Instrument Assisted Soft Tissue Mobilization (Experimental): In the application group, Instrument Assisted Soft Tissue Mobilization will be applied to the Trapezius and Sternocleideomastoideus muscles for 90 seconds.
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization
- Sham Instrument Assisted Soft Tissue Mobilization (Sham Comparator): In the sham application group, 90 degrees to 90 seconds will be applied to the Trapezius and Sternocleideomastoideus muscles without applying pressure.
  Interventions: Other: Sham
- Control (No Intervention): No application will be made to the control group.

INTERVENTIONS:
Other: Instrument Assisted Soft Tissue Mobilization — Bilateral Instrument assisted soft tissue mobilization application will be applied in a single session to the trapezius and sternocleideomastoideus muscles.
  Arms: Instrument Assisted Soft Tissue Mobilization
Other: Sham — Bilateral sham Instrument assisted soft tissue mobilization application will be applied in a single session to the trapezius and sternocleideomastoideus muscles.
  Arms: Sham Instrument Assisted Soft Tissue Mobilization

SUMMARY:
Chronic neck pain causes errors in joint position. There are studies in the literature suggesting that the application of instrument-assisted soft tissue mobilization improves the sense of joint position. There are no studies that acutely examine this practice on joint position sense and pain in the cervical region. As a result of our study, we will investigate the effects of instrument-assisted soft tissue mobilization in a single session on perception of pain and joint position.

ELIGIBILITY:
Inclusion Criteria:

* • Being diagnosed with chronic neck pain,

  * To be in the age range of 18-65.

Exclusion Criteria:

* • Those taking any analgesic medication

  * Those with acute injury or infection,
  * Those with open wounds, Osteoporosis,
  * Broken,
  * Hematoma, Those with acute cardiac, liver and kidney problems,
  * Those with connective tissue disease, Rheumatoid arthritis, osteoarthritis, Cancer,
  * Those with circulation problems,
  * Those with peripheral vascular disease, Epilepsy, Surgery history in the cervical area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-06-26 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Cervical Pain at 2 minutes | Baseline and 2 minutes after intervention
  Pain will be evaluated with Visual Analog Scale.
Change from Baseline Joint Position Sense at 2 minutes | Baseline and 2 minutes after intervention
  Joint Position Sense will be evaluated Cervical Range of Motion Device

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gercek H, Unuvar BS, Umit Yemisci O, Aytar A. Acute effects of instrument assisted soft tissue mobilization technique on pain and joint position error in individuals with chronic neck pain: a double-blind, randomized controlled trial. Somatosens Mot Res. 2023 Mar;40(1):25-32. doi: 10.1080/08990220.2022.2157388. Epub 2022 Dec 20. PMID 36538383